CLINICAL TRIAL: NCT04188522
Title: Imaging the Network: Using MEG to Determine the Pathophysiology Underlying Post-Stroke Cognitive Impairment
Brief Title: Imaging Post-Stroke Recovery: Using MEG to Evaluate Cognition
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland, College Park (Other); American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00122221; 18IPA34170313 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Stroke Sequelae; Stroke/Brain Attack
MeSH Terms: conditions — Stroke | interventions — Magnetoencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minor Stroke: We will enroll a cohort of 15 adult patients previously admitted to Johns Hopkins Bayview Medical Center with small/minor acute ischemic stroke visible on neuroimaging. Patients will follow-up in clinic 4-6 weeks following hospital discharge. To be eligible for the study, patients must have a "minor stroke", defined as NIH Stroke Scale score at follow-up of less than or equal to 8, modified Rankin score of 0-2, be competent speakers of English, and have no prior history of stroke, dementia, or untreated psychiatric disease. Those with proximal large vessel (M1) or branch (M2) occlusions will be excluded.
  *Based on preliminary results we have expanded our trial and will continue to recruit up to 40 patients with minor stroke.
  Interventions: Diagnostic Test: Magnetoencephalography (MEG)
- Controls: For comparison, we will recruit a group of age-similar controls (n=15) without neurologic disease or prior clinical history of stroke.
  Interventions: Diagnostic Test: Magnetoencephalography (MEG)

INTERVENTIONS:
Diagnostic Test: Magnetoencephalography (MEG) — Participants will undergo MEG at the University of Maryland (College Park) to measure cerebral activity while performing a visual naming task. The Montreal Cognitive Assessment (MOCA) will also be administered.
  Other Names: Cognitive Testing

SUMMARY:
This is a study using magnetoencephalography (MEG) to look at recovery in those with minor stroke. The investigators know that these individuals report difficulties in attention, concentration, multi-tasking, energy level, and processing speed that appear to be independent of lesion size or location. The underlying pathophysiology is unclear; however, anecdotally, many individuals are significantly improved by 6 months post-stroke. One hypothesis is that a single lesion, regardless of size, may disrupt the classic neural networks required for cognitive function. The investigators are currently collecting data to better characterize these difficulties and stroke patients' recovery as part of a previously approved recovery study. In this sub-study, the investigators propose to add MEG at 1 and 6 months in a subset of individuals with small: 1) subcortical, and 2) cortical lesions. The investigators will partner with colleagues at the University of Maryland (College Park), who are well experienced with MEG to conduct this research. In addition a control population of age-similar individuals will be recruited for comparison. Cerebral activation patterns of individuals with stroke versus controls will be compared, both across patients with stroke at a given time point, and within subjects from 1 to 6 months to determine the association of abnormal activation with cognitive dysfunction and recovery.

**The investigators have recently extended follow-up by adding an additional assessment at 12 months and will enroll additional participants (up to 40 patients with minor stroke, 15 age-similar controls).

DETAILED DESCRIPTION:
This is a prospective longitudinal study of patients with minor stroke versus age-similar controls that will make use of the following protocol:

* Patients are admitted to the hospital for acute stroke and undergo work-up including MRI; they are entered into a clinical outcomes database (routine clinical care)
* All patients are scheduled for an appointment in the Bayview Stroke Intervention Clinic approximately 4-6 weeks +/- 4 weeks post-stroke
* Seen at 4-6 weeks (routine care)- consented and tested if enrolled (per research protocol, as part of a prior approved study on stroke recovery)
* Those meeting inclusion criteria for MEG testing will be consented and undergo the following additional procedures: 1 month MEG visit at the University of Maryland- brain activity will be measured at rest and during cognitive tasks evaluating domains such as: executive function, attention, and multi-tasking including a visual naming test Repeat MEG at approximately 6 months +/- 4 weeks post-stroke

University of Maryland's MEG Protocol:

The head shape will be measured using a 3D tracking system. This involves using a plastic stylus to mark a series of points around the head that will map the entire surface of the head. In addition, each of three "fiducial" points; one in front of each ear and one above and between the eyes will be marked. The purpose of the head shape measurement is to be able to co-localize brain activity recorded with the MEG with the subject's MRI.

Magnetic fields will be recorded using a 275-channel whole-head MEG system. A third-order gradient will be used for noise cancellation.

The MEG system non- invasively measures the magnetoencephalographic (MEG) signals (and, optionally, electroencephalographic EEG signals) produced by electrically active tissue of the brain. These signals are recorded by a computerized data acquisition system, displayed, and may then be interpreted by trained physicians to help localize these active areas. The location may then be correlated with anatomical information of the brain. MEG is routinely used to identify the locations of visual, auditory, somatosensory, and motor cortex in the brain. MEG is also used to non-invasively locate regions of epileptic activity within the brain. The localization information provided by MEG may be used, in conjunction with other diagnostic data, in neurosurgical planning.

The total length of the MEG recordings will depend on the length of the tasks (an estimate of 30-45 min has been used). There will be a 2-5 -minute break between each run. For all runs magnetic fields will be recorded in 42 consecutive 10-second trials. In this way if there are artifacts during the session, such as the subject moving his or her head, the 10-second trial during which this occurs can be eliminated from analysis.

Patients will return for their 6 month and 12 month post-stroke follow-up appointments (routine care) and testing (if part of the recovery study).

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) admitted to Bayview Medical Center Neurology.
2. Evidence of acute ischemic stroke (CT or MRI)- lacunar stroke or branch occlusion (M3/A3/P3 or smaller) OR NIHSS ≤ 8 on admission.
3. Competent speaker of English (by self or family report) prior to stroke.
4. Return for follow-up 4-6 weeks post event (+/- 4 wks).
5. Cognitive deficits present on initial testing.** unique to MEG study
6. Willing to travel to the University of Maryland twice for MEG.** unique to MEG study
7. Fully independent functionally and able to travel to the University of Maryland unassisted.** unique to MEG study

Exclusion Criteria:

1. Primary intracerebral hemorrhage- as evidenced by blood on head CT or MRI.
2. Previous neurological disease (e.g., dementia, multiple sclerosis, prior symptomatic stroke). Incidental asymptomatic lacunar strokes found on imaging will not be excluded as prior disease.
3. Uncorrected hearing or visual loss.
4. Large vessel occlusion.
5. Presence of any of the following that would lead to significant artifact on MEG: cardiac pacemaker, intracranial clips, metal implants, or external clips within 10mm of the head, metal in the eyes.** unique to MEG study
6. Claustrophobia, obesity, and/or any other reason leading to difficulty staying in the MEG for up to 1 hour.** unique to MEG study
7. For controls- clinical history of stroke or other neurological dysfunction (seizure, multiple sclerosis, etc.); psychiatric disease

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from those recently hospitalized with minor stroke at Johns Hopkins Bayview Medical Center (see inclusion criteria).
  Controls will include friends, family, and other volunteers of similar age meeting Inclusion Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cerebral Activity Measured Using Magnetoencephalography (MEG) | Up to 10 weeks
  Global patterns of cerebral activity as well as individual brain areas important for cognitive processing will be analyzed for differences with respect to amplitude, latency, and frequency.
Cerebral Activity Measured Using Magnetoencephalography (MEG) | Up to 6 months
  Global patterns of cerebral activity as well as individual brain areas important for cognitive processing will be analyzed for differences with respect to amplitude, latency, and frequency.
Cerebral Activity Measured Using Magnetoencephalography (MEG) | Up to 12 months
  Global patterns of cerebral activity as well as individual brain areas important for cognitive processing will be analyzed for differences with respect to amplitude, latency, and frequency.
Reaction Time | Up to 10 weeks
  Reaction times will be recorded and compared during the visual naming task
Reaction Time | Up to 6 months
  Reaction times will be recorded and compared during the visual naming task
Reaction Time | Up to 12 months
  Reaction times will be recorded and compared during the visual naming task

SECONDARY OUTCOMES:
MOCA | Up to 10 weeks
  Scores on the MOCA will be compared between those with minor stroke and controls
MOCA | Up to 6 months
  Scores on the MOCA will be compared between those with minor stroke and controls
MOCA | Up to 12 months
  Scores on the MOCA will be compared between those with minor stroke and controls

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth B Marsh, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available upon request of the PI. Otherwise, de-identified results will be reported in aggregate.
Supporting Information: Study Protocol, SAP
Time Frame: Complete results will be published at the conclusion of the study, though initial results are published and available for review (final citation below).
Access Criteria: Upon request. In addition, anonymized MEG fif files used for preliminary analysis and publication have been deposited in the University of Maryland Data Repositories. All other data pertaining to the published study are included in the article and Supporting Information (SI) Appendix.
URL: https://doi.org/10.13016/n9j1-mwne

REFERENCES:
- [Background] Chen K, Marsh EB. Chronic post-stroke fatigue: It may no longer be about the stroke itself. Clin Neurol Neurosurg. 2018 Nov;174:192-197. doi: 10.1016/j.clineuro.2018.09.027. Epub 2018 Sep 17. PMID 30266010
- [Background] Marsh EB, Lawrence E, Gottesman RF, Llinas RH. The NIH Stroke Scale Has Limited Utility in Accurate Daily Monitoring of Neurologic Status. Neurohospitalist. 2016 Jul;6(3):97-101. doi: 10.1177/1941874415619964. Epub 2015 Dec 13. PMID 27366291
- [Background] Marsh EB, Lawrence E, Hillis AE, Chen K, Gottesman RF, Llinas RH. Pre-stroke employment results in better patient-reported outcomes after minor stroke: Short title: Functional outcomes after minor stroke. Clin Neurol Neurosurg. 2018 Feb;165:38-42. doi: 10.1016/j.clineuro.2017.12.020. Epub 2017 Dec 27. PMID 29306185
- [Result] Marsh EB, Brodbeck C, Llinas RH, Mallick D, Kulasingham JP, Simon JZ, Llinas RR. Poststroke acute dysexecutive syndrome, a disorder resulting from minor stroke due to disruption of network dynamics. Proc Natl Acad Sci U S A. 2020 Dec 29;117(52):33578-33585. doi: 10.1073/pnas.2013231117. Epub 2020 Dec 14. PMID 33318200
- See also: Marsh Lab Website — http://marshlab.org